CLINICAL TRIAL: NCT06259487
Title: Study on the Impact of Coordinated Immunizations Against RSV and Influenza on the Prognosis in Patients With Chronic Heart Failure.
Brief Title: Coordinated Vaccination Against RSV and Influenza in Patients With Chronic Heart Failure and Its Impact on Prognosis.
Acronym: VACCINE-CHF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Jan Biegus, MD, PhD, MD, PhD, Wroclaw Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 325/2023N
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure; RSV Infection; Influenza; Vaccines
Keywords: heart failure; RSV; Influenza; Vaccination; Immunization; Prognosis
MeSH Terms: conditions — Heart Failure; Respiratory Syncytial Virus Infections; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coordinated Vaccination against RSV and Influenza (Experimental): Patients receiving vaccinations against Respiratory Syncytial Virus (RSV) and influenza provided by the research team (i.e. during cardiology visits).
  Interventions: Biological: Coordinated Vaccination
- Standard of care (Active Comparator): Patients following standard recommendations for protective vaccinations (i.e., receiving vaccinations at vaccination points).
  Interventions: Behavioral: Following recommendations

INTERVENTIONS:
Biological: Coordinated Vaccination — Coordinated Vaccination against Respiratory Syncytial Virus (RSV) and influenza provided by the research team (i.e., during cardiology visits)
  Arms: Coordinated Vaccination against RSV and Influenza
Behavioral: Following recommendations — Guidance on following the standard recommendations for protective vaccinations (i.e., receiving vaccinations at vaccination points).
  Arms: Standard of care

SUMMARY:
This prospective, single-centre, open-label, randomized study aims to determine whether coordinated care in administering protective vaccinations (against Respiratory Syncytial Virus (RSV) and influenza) impacts the prognosis of patients with chronic heart failure.

The main question it aims to answer is:

• Does coordinated care through vaccinations improve the prognosis of patients with chronic heart failure?

DETAILED DESCRIPTION:
The study aims to determine whether coordinated care in the form of administering protective vaccinations affects the prognosis of patients with chronic heart failure. The study will involve analyzing epidemiological data for each participant, followed by randomization into two treatment paths: receiving vaccinations against Respiratory Syncytial Virus (RSV) and influenza provided by the research team (i.e., during cardiology visits) versus following standard recommendations for protective vaccinations (i.e., receiving vaccinations at vaccination points). All vaccinations will be administered using vaccines registered with the appropriate authorities and approved for use in the EU and Poland.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Willingness to provide informed consent for participation in the study
* Diagnosis of heart failure
* No previous vaccination against RSV or influenza

Exclusion Criteria:

* History of an anaphylactic reaction to vaccination
* Hypersensitivity to any component of the vaccine
* Receipt of vaccination against RSV or influenza in the current infectious
* Active infection
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint: All-cause mortality, hospitalization due to heart failure, and the clinical signs of infection, characterized by a body temperature exceeding 38 degrees Celsius. | 180 days
  Number of days from the intervention to the occurrence of the composite endpoint.

CONTACTS AND LOCATIONS:
Locations (1):
- Wroclaw Medical University, Wroclaw, Dolnyslask, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biegus J, Szenborn L, Zymlinski R, Zakliczynski M, Reczuch K, Guzik M, Urban S, Rosiek-Biegus M, Jankowiak B, Iwanek G, Fudim M, Ponikowski P. The early safety profile of simultaneous vaccination against influenza and Respiratory Syncytial Virus (RSV) in patients with high-risk heart failure. Vaccine. 2024 Apr 30;42(12):2937-2940. doi: 10.1016/j.vaccine.2024.03.060. Epub 2024 Mar 25. PMID 38531725